CLINICAL TRIAL: NCT01865981
Title: Cellular Reprogramming as a Tool to Characterise the Cellular Electrophysiology of Familial Arrhythmia
Brief Title: Investigating Hereditary Cardiac Disease by Reprogramming Skin Cells to Heart Muscle
Acronym: CLUE
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: 2012CA04; T13/21 (Other Grant/Funding Number: Tenovus Tayside)
Record Dates: First submitted 2013-05-15; First posted 2013-05-31 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Eletrophysiology of iPS-derived Cardiomyocytes
Keywords: iPS cells; cardiomyocytes; Brugada; Ventricular Fibrillation; electrophysiology
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: None Retained — Skin biopsies will be extracted and used to derive fibroblasts. These will be retained and reprogrammed to iPS cells (also to be retained). Derived cell lines are not considered a tissue under the UK Human Tissue Act
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hereditary VF: Patients with hereditary ventricular fibrillation, negative for known mutations
- Brugada: Patients suffering from Brugada syndrome

SUMMARY:
Hereditary cardiac arrhythmias (genetically caused disturbances of heart rhythm) are life threatening conditions affecting otherwise healthy young individuals. Due to the inaccessibility of heart tissue, the abnormal electrical current(s) in the heart cells causing the rhythm disturbance can be difficult to study in detail and therefore in many cases remain untreatable. The investigators propose to study heart cell electrical function from such patients by reprogramming skin cells to become stem cells and then differentiating them to heart muscle cells.

The hypothesis of the study is that the differentiated cardiac cells will display electrical abnormalities dependent on the mutation causing the disease. These abnormalities can therefore provide a clue as to the nature of the mutation causing the disease or information about its effective management

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of Brugada Syndrome (ECG findings)
* mutation positive or mutation negative
* Idiopathic ventricular fibrillation

Exclusion Criteria:

* not able to give informed consent
* Age less than 18 years
* clinical diagnosis ambiguous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arrhythmic patients participating in the Familial Arrhythmia Network Scotland (FANS)
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Derivation of iPS cells | 12 months
  Induced pluripotent cells will be derived from all participants in the study. Differences in the efficiency of iPS cell generation from different patients will be recorded, and correlated with disease status and age. iPS cell generation will be confirmed by pluripotency markers (stable endogenous gene expression of Nanog, Oct4, Sox2; colony formation; expression of SSEA4) and ability to differentiate in the absence of self-renewal stimulus (ability to self-renew in the absence of self-renewal stimulus -loss of markers above)

SECONDARY OUTCOMES:
Differentiation of iPS cells to cardiomyocytes | 12 months
  The ability of each iPS cell line to differentiate into spontaneously beating cardiomyocytes will be assessed. Efficiency of differentiation per lina and per patient will be recorded.
Electrophysiology on iPS-derived cardiomyocytes | 12 months
  Ability to collect electrophysiological measurements from iPS-derived cardiomyocytes will be asssessed. Resting membrane potential, Ca2+, K+ current function and sponteneous and induced depolarisation will be measured per line and per patient. Correlations with patient disease phenotype will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marios P Stavridis, PhD, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, Angus, United Kingdom